CLINICAL TRIAL: NCT05762549
Title: Prevalenza Dell'Ipercortisolismo Occulto Nell'Osteoporosi
Brief Title: Prevalence of Hidden Hypercortisolism in Osteoporosis
Acronym: OSTCOR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 05L101
Record Dates: First submitted 2023-02-26; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Osteoporosis; Cortisol Excess
MeSH Terms: conditions — Osteoporosis; ACTH Syndrome, Ectopic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goals of this observational study are the following:

i) to assess the prevalence of hidden hypercortisolism (HidHyCo) in a sample of osteoporotic patients; ii) to compare the clinical characteristics between osteoporotic/osteopenic patients with HidHyCo and those without HidHyCo in order to determine the clinical characteristics more frequently associated with the HidHyCo presence in the osteoporotic population and to identify those osteoporotic patients worthy of HidHyCo screening.

In all patients who have been included in the study and who have given the informed consent to participate in the study we will perform 1 mg overnight dexamethasone suppression test (F-1mgDST).

In all subjects with F-1mgDST >1.8 mcg/dL, cortisol levels after two-day low dose (2 mg/day) dexamethasone suppression test (F-2mgx2dDST) will be measured.

Patients with F-2mgx2dDST above >1.8 mcg/dL will be considered affected with HidHyCo and will be managed following the available guidelines for hypercortisolism.

The HidHyCo could be present in a not negligible percentage of osteopenic/osteoporotic patients. In these patients, osteoporosis and, if present, other comorbidities (i.e. hypertension and/or diabetes) can improve by the surgical resection of the adrenal or pituitary adenoma if feasible, or by the use of drugs able to modulate cortisol secretion or glucocorticoid sensitivity.

DETAILED DESCRIPTION:
Clinically overt hypercortisolism (i.e. Cushing's syndrome) leads to hypertension, central obesity, diabetes and osteoporosis.

More recently, even the condition of mild and asymptomatic hypercortisolism has been associated with increased prevalence of chronic complications of cortisol excess and mortality. In patients with osteoporosis this form of hypercortisolism may remain occult (hidden hypercortisolism, HidHyCo), until its presence is suspected on the basis of particular characteristics of the underlying disease.

By definition, HidHyCo is a condition of cortisol excess in the absence of its classical signs and symptoms. Although asymptomatic, however, this subtle cortisol excess is associated with an increased risk of osteoporosis and fragility fractures.

Moreover, HidHyCo prevalence seems to be increased in osteoporotic patients. In particular, the prevalence of HidHyCo in patients with low bone mineral density and with fragility fracture has been reported to be 1.7-9.9% and 1.9-17.6%, respectively.

The HidHyCo case finding is of utmost importance since these patients experience an impressive reduction of the fracture risk after the normalization of cortisol levels. However, given the high prevalence of bone fragility and the relatively low diagnostic accuracy of the currently available tests for the HidHyCo detection, a mass screening for HidHyCo is considered unthinkable. Therefore, the issue of which osteoporotic patient has to be screened for HidHyCo has recently become a widely debated topic, but as now, no guidelines are available for addressing the HidHyCo screening in osteoporosis.

Therefore, the aims of the present study protocol are the following: i) to assess the HidHyCo prevalence in a sample of osteoporotic patients; ii) to compare the clinical characteristics between osteoporotic/osteopenic patients with HidHyCo and those without HidHyCo in order to determine the clinical characteristics more frequently associated with the HidHyCo presence in the osteoporotic population and to identify those osteoporotic patients worthy of HidHyCo screening.

In all patients who have been included in the study and who have given the informed consent to participate in the study the following vital and anthropometric parameters will be recorded: blood pressure, heart rate, weight, height, body mass index (BMI), abdominal circumference and waist-to-hip ratio. Moreover, the following variables will be collected: familiar history of fragility fracture, smoking habit, main comorbidities, history of falls, previous clinical fragility fractures, ongoing pharmacological treatment (in particular type and number of antihypertensive, lipid lowering, anti-diabetic and anti-osteoporotic drugs), previous anti-osteoporotic treatments, in females regularity of menses or age of menopause and in males testosterone levels. Questionnaires for assessing daily calcium intake and physical activity will be administered to all patients.

At the time of enrolment, the results of first tier investigations according to national guidelines (i.e. serum erythrocyte sedimentation rate, complete blood count, serum protein electrophoresis, serum calcium levels, serum phosphate levels, total alkaline phosphatase, serum creatinine, 24-h urinary calcium) will be also registered. Moreover, other calcium-phosphate metabolism parameters (i.e. serum ionized calcium, serum parathyroid hormone, serum 25-OH-vitamin D, serum ß-CrossLaps, bone alkaline phosphatase) and routine determinations (i.e. fasting glucose, insulin, glycated haemoglobin, total cholesterol, low density lipoprotein, high density lipoprotein, triglycerides, transaminases) will be recorded, if available.

According to the good clinical practice, in all patients bone mineral density will be assessed by dual-energy X-ray Absorptiometry (Hologic or Lunar bone densitometers) and the presence of asymptomatic vertebral fractures will be checked by conventional spinal radiographs using the semi-quantitative visual assessment described by Genant et al., defined as a reduction of >20% in anterior, middle, or posterior vertebral height.

Finally, iIn all patients who have been included in the study and who have given the informed consent to participate in the study we will perform 1 mg overnight dexamethasone suppression test (F-1mgDST). In all subjects with F-1mgDST >1.8 mcg/dL, cortisol levels after two-day low dose (2 mg/day) dexamethasone suppression test (F-2mgx2dDST) will be measured.

Patients with F-2mgx2dDST above >1.8 mcg/dL will be considered affected with HidHyCo and will be managed following the available guidelines for hypercortisolism.

The HidHyCo prevalence in osteopenic/osteoporotic patients and its 95% interval confidence will be calculated.Then, we will compare the clinical and biochemical characteristics of osteoporotic/osteopenic patients with HidHyCo and those without HidHyCo.

The sample size has been calculated in order to have an adequate number of HidHyCo cases to determine the characteristics of osteoporotic patients suggestive for the presence of HidHyCo. Since HidHyCo may be estimated to have at least a 3% prevalence in osteoporotic patients, a sample of 1500 osteoporotic patients should be adequate to find no less than 45 HidHyCo cases.

Indeed, based on preliminary data, it is possible to assume that HidHyCo is present in a not negligible percentage of osteopenic/osteoporotic patients.

The presence of osteoporosis associated with a poorly controlled hypertension and/or diabetes or with a history of cardiovascular events (osteopenia with comorbidities) or the presence of fragility fractures in the presence of not osteoporotic bone density, in an eugonadal state and/or on osteoporotic treatment with bone-active drugs may be the variables potentially associated with an increased probability of having HidHyCo.

By testing our sample of osteoporotic patients for HidHyCo, we aim at obtaining information regarding the pre-test probability of a single individual of having a subtle cortisol excess and, if feasible, at developing a clinical model for the identification in outpatient osteoporosis clinics of subjects worthy of HidHyCo testing, thus avoiding a mass screening.

In HidHyCo patients, osteoporosis and, if present, other comorbidities (i.e. hypertension and/or diabetes) can improve by the surgical resection of the adrenal or pituitary adenoma if feasible, or by the use of drugs able to modulate cortisol secretion or glucocorticoid sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* presence of osteoporosis (i.e. lumbar and/or femoral BMD T-score < -2.5 and/or Z-score < -2.0 and/or fragility fracture of hip, spine, wrist, humerus, malleolus or ribs);
* presence of osteopenia (i.e. lumbar and/or femoral BMD T-score between -1.0 and -2.5) in addition to hypertension treated with at least 2 drugs or not well controlled hypertension (sustained blood pressure above 150/100 mmHg) and/or diabetes and/or to a history of cardiovascular events (such as deep vein thrombosis, coronary heart disease, myocardial infarction, stroke).

Exclusion Criteria:

* pregnancy/breastfeeding, sleep apnea, prepuberal onset of hypertension, hormonal hypersecreting adrenal mass, signs/symptoms of hypercortisolism;
* already known secondary osteoporosis with the exception of hypercalciuria;
* drugs influencing the bone metabolism with the exception of diuretics, anti-diabetics and anticoagulants;
* conditions associated with increased hypothalamic-pituitary-adrenal (HPA) axis activity, severe autoimmune/rheumatologic and hematologic diseases, alcoholism, chronic kidney disease (glomerular filtration rate <60 ml/min);
* drugs influencing the HPA axis activity or the dexamethasone metabolism.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals referred to our outpatients clinics for osteoporosis
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-05-26 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of hidden hypercortisolism in patients with osteoporosis or osteopenia plus the comorbidities possibly associated with cortisol excess | 18 months
  To evaluate the prevalence of hidden hypercortisolism in patients with osteoporosis or osteopenia plus the comorbidities possibly associated with cortisol excess.

SECONDARY OUTCOMES:
Predictors of the presence of HidHyCo in in patients with osteoporosis or osteopenia associated with comorbidities. | 18 months
  To evaluate the characteristics predictive of the presence of HidHyCo in in patients with osteoporosis or osteopenia associated with comorbidities.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Cairoli, MD, Principal Investigator — Istituto Auxologico Italiano
Locations (5):
- Italy (5):
  - U.O.C. Medicina Interna, Azienda Ospedaliero Universitaria Policlinico "G. Rodolico - San Marco", Catania
  - U.O.C. Endocrinologia, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - U.O.S. Endocrinologia, Ospedale "Casa Sollievo della Sofferenza" IRCCS, San Giovanni Rotondo
  - Dipartimento di Scienze Mediche, Chirurgiche e Neuroscienze, Azienda Ospedaliero-Universitaria Senese di Santa Maria alle Scotte, Siena
  - S.O.C. Endocrinologia e Malattie del Metabolismo, Presidio Ospedaliero Universitario "Santa Maria della Misericordia", Azienda Sanitaria-Universitaria Friuli Centrale, Udine